CLINICAL TRIAL: NCT04072016
Title: The Beacon Study: A Prospective, Multicenter Study to Evaluate the Safety and Effectiveness of Beacon Aqueous Microshunt for Refractory Glaucoma
Brief Title: Study of the Beacon Aqueous Microshunt in Patients With Refractory Glaucoma
Acronym: Beacon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant risks (e.g., infection, endothelial cell loss) and high rate of channel plugging associated with product use.
Sponsor: MicroOptx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4046
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Beacon Aqueous Microshunt (Experimental)
  Interventions: Device: Beacon Aqueous Microshunt

INTERVENTIONS:
Device: Beacon Aqueous Microshunt — The Beacon Aqueous Microshunt (BAM) is an implantable device intended to reduce intraocular pressure (IOP) in patients with refractory glaucoma by shunting aqueous humor from the anterior chamber to the surface of the eye.

SUMMARY:
This is a prospective, multicenter, single-arm clinical study to evaluate the safety and effectiveness of Beacon Aqueous Microshunt in patients with refractory glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-85 years.
2. Refractory glaucoma: Prior failure of filtering/cilioablative procedure and/or uncontrolled IOP on maximum-tolerated medication (i.e. >=4 classes of topical lowering medications, or fewer in the case of tolerability or efficacy issues).
3. Primary open-angle, traumatic or neovascular glaucoma.
4. Medicated DIOP ≥20 mmHg and ≤45 mmHg on maximum-tolerated medical therapy. Note: No washout; medications stabilized 30 days prior to assessment.
5. Baseline BCVA of light perception or better in study eye.
6. Visual field defects consistent with glaucomatous optic nerve damage.
7. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   * Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage;
   * Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or
   * Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue 8. Visual field mean deviation (MD) by Humphrey Visual Field: Visual field defects consistent with glaucomatous optic nerve damage and mean deviation worse than -3 dB in the study eye; and at least one of the following two findings:
   * A cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level on the pattern deviation (PD) plot; and/or
   * Glaucoma hemi-field test "outside normal limits".

9. At least two contiguous clock hours of intact conjunctiva near the limbus between clock hours of 9:00 and 03:00 in the study eye.

10. Adequate space in the anterior chamber by Spaeth Grade C, D or E for iris insertion (with indentation).

11. Participant has the understanding, ability, and willingness to fully comply with study procedures and postoperative care instructions.

12. Participant understands and signs the informed consent.

Exclusion Criteria:

1. No light perception vision.
2. Conditions of active neovascular conditions, such as active iris or corneal neovascularization, or active proliferative retinopathy in study eye.
3. Pigmentary glaucoma in study eye.
4. Pseudoexfoliation syndrome in study eye.
5. Angle-closure glaucoma in study eye.
6. Iridocorneal endothelial syndrome in study eye.
7. Uveitic glaucoma in the study eye.
8. Epithelial or fibrous downgrowth in the study eye.
9. Best corrected visual acuity (BCVA) worse than 20/200 in the non-study eye.
10. Corneal conditions in study eye inhibiting normal incisional healing (e.g. Fuch's dystrophy) or impair visualization of implant inside the anterior chamber.
11. Prior intraocular surgery in study eye within ≤6 months before the preoperative visit (including phacoemulsification).
12. Central corneal endothelial cell count of less than 1600 cells/mm2 in the study eye.
13. Anticipated need for ocular surgery or retinal laser procedure in the study eye within the 12-month follow-up period.
14. Need for glaucoma surgery combined with other ocular procedures in the study eye at time of implant (e.g. cataract surgery, penetrating keratoplasty, or retinal surgery).
15. Unwilling to discontinue contact lens use in the study eye after surgery.
16. Central corneal thickness ≤490μm or ≥620μm.
17. Clinically significant inflammation or infection in the study eye within 60 days prior to the preoperative visit (e.g., blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection) or any systemic infection. For purposes of this study, clinically significant is considered any such condition requiring prescription therapy.
18. Any condition that prevents the device implantation in the superior region of the study eye.
19. Vitreous in the anterior chamber for which a vitrectomy is anticipated.
20. Functionally significant cataract in the study eye.
21. Other clinical conditions:

    1. Poorly controlled diabetes (Type I or Type II) as determined by HbA1c >8 within 3 months of implant.
    2. Cancer requiring treatment during the duration of the study.
    3. Any drugs (e.g.: immunosuppressive drugs) or co-morbidity that might inhibit wound healing.
22. Participation in any other clinical study during participation in this study.
23. Engage in activities that involve submerging their head under water, such as diving or swimming.
24. Women who are (i) pregnant, (ii) nursing, (iii) planning a pregnancy and (iv) of childbearing potential not using a reliable method of contraception.
25. Life expectancy <1 year.

If both eyes are eligible, the eye with the worse BCVA will be selected.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness via Intraocular Pressure Reduction | 12 Months
  20% mean diurnal IOP reduction from baseline, on the same number or fewer topical IOP-lowering medications
Safety via Serious and Adverse Event Reporting | 12 Months
  Rate of occurrence of serious procedure-related and/or device-related adverse events.

SECONDARY OUTCOMES:
Responder rate defined as achieving at least 20% mean diurnal IOP reduction from baseline | 12 Months
Mean Change from baseline in IOP | 12 Months
Schirmer tear test - Mean change from baseline | 12 Months
Proportion of Eyes Achieving Specific IOP Targets (≤18 mmHg, ≤17 mmHg, ≤16 mmHg, ≤15 mmHg, ≤14 mmHg, ≤13 mmHg, and ≤12 mmHg) compared to baseline | 12 Months
Number of topical IOP-lowering medications - Mean change from baseline | 12 Months
Kaplan-Meier Analysis of Failure | 12 Months
  Glaucoma-related secondary surgical intervention with or without device explant, device explant alone, or not achieving >20% IOP reduction on the same number of medications or fewer
Rate of ocular and non-ocular adverse events | 12 Months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Icon Eye Care, Grand Junction, Colorado
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - iWorks Laser and Vision Center, Dayton, Ohio
- Institut de l'oeil des Laurentides, Boisbriand, Qubec, Canada